CLINICAL TRIAL: NCT02284555
Title: A Single Centre, Open, Non-controlled Study in Healthy Subjects to Assess the Eradication of Nasal Carriage of Staphylococcus Aureus (SA) Following a Five Day Course of Mupirocin (Bactroban 2% Nasal Ointment) Using a Broth Enriched Culture Microbiological Assessment.
Brief Title: Study to Assess Eradication of Nasal Carriage of Staphylococcus Aureus (SA) With Mupirocin (Bactroban 2% Nasal Ointment)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Destiny Pharma Plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XF-MupC01
Record Dates: First submitted 2014-10-21; First posted 2014-11-06 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Staphylococcal Infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mupirocin 2% nasal Ointment (Experimental): Mupirocin (Bactroban 2% nasal ointment) will be administered twice daily for 5 days in accordance with the Summary of Product Characteristics (SmPC).
  Interventions: Drug: Mupirocin

INTERVENTIONS:
Drug: Mupirocin — Mupirocin (Bactroban 2% Nasal Ointment) will be administered twice daily for five days in accordance with the SmPC.
  Other Names: Bactroban

SUMMARY:
This study will assess the nasal eradication of SA in healthy subjects following treatment with mupirocin 2% (Bactroban 2% Nasal Ointment) twice daily for 5 days, by means of a broth enriched culture microbial assay. The sensitivities of broth enrichment and plating assay methods will be compared. The safety and tolerability of Bactroban 2% Nasal Ointment will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy male or female subjects aged between 18 and 75 years.
2. Subjects confirmed to be persistent nasal SA carriers, defined by 3 separate, SA positive cultures from nasal swabs. Two positive cultures should be obtained at screening visits up to 12 weeks prior to inclusion and at least two weeks apart. The final confirmatory culture should be obtained from a baseline nasal swab prior to administration of the first dose.
3. Subjects who are able and willing to provide written informed consent to participate in the study
4. Subjects who have a body mass index (BMI) ≥18.5 kg/m2 and ≤ 32 kg/m2.
5. Subjects who agree not to take part in another clinical trial at any time during the study period.

Exclusion Criteria:

1. Female subjects who are or may be pregnant or who are lactating.
2. Subjects who have any acute or chronic illness or infection.
3. Subjects who have smoked within the 3 months prior to screening (confirmed by urinary cotinine test).
4. Subjects who are females of child-bearing potential, defined as being physiologically capable of becoming pregnant, UNLESS using one or more of the following acceptable methods of contraception; established use of oral, injected or implanted hormonal contraception, intrauterine Device (IUD or Coil AND barrier Method (condom or diaphragm or cervical/vault cap) plus spermicidal cream/gel. Contraceptive use should continue throughout the study and for 1 month following completion of the study.
5. Subjects who are fertile males, defined as all males physiologically capable of conceiving offspring, UNLESS the subject agrees to comply with acceptable contraception e.g. condom plus spermicidal cream/gel. Contraceptive use should continue throughout the study and for 3 months following completion of the study.
6. Subject with any open wound, lesion, inflammation, erythema or infection affecting the nostrils, nose, upper lip and area of skin close to the nose. This includes herpes simplex lesions and discoid lupus.
7. Subjects who have a currently symptomatic upper respiratory tract infection, nasopharyngitis, influenza or condition involving increase in nasal secretion such as seasonal or chronic, allergic rhinitis.
8. Subjects with a history of drug or alcohol abuse in the previous 12 months or who have a positive urine drug test for substances of abuse.
9. Subjects with a known clinically significant history of atopy or hypersensitivity to any drug or latex.
10. Subjects with a history of serious illness, cancer or psychiatric condition.
11. Subjects who have been treated with or have taken any prescribed or over-the-counter medication within the previous 14 days, with the exception of hormonal contraceptives or hormone replacement therapy.
12. Subjects who have taken or used topical or systemic antibiotics within the month prior to screening.
13. Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for human immunodeficiency virus (HIV) antibodies
14. Subjects who have participated in a clinical trial within the last 3 months.
15. Subjects with any clinically significant abnormality in vital signs or laboratory analyses at screening or at baseline, based on the opinion of the investigator.
16. Subjects with nasal polyps or significant anatomical nasal abnormality.
17. Subjects with a history of nasal surgery, including cauterization in the last 12 months.
18. Subjects with a history of multiple episodes [>3] of epistaxis within the last 12 months.
19. Subjects with in-situ nasal jewellery or open nasal piercings.
20. Subjects with a history of abnormal bleeding, bruising, frequent nosebleeds or a diagnosis of von Willebrand disease.
21. Subjects who have or have had an autoimmune disease.
22. Subjects with hypersensitivity to any of the ingredients of Bactroban® Nasal Ointment i.e. mupirocin, white soft paraffin, Softisan 649 (mixed diglycerinester of fatty acids).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Mr Hayter, BSc, Study Director — Destiny Pharma Plc
Locations (1):
- Simbec Reseach Ltd, Wales, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mupirocin 2% Nasal Ointment
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mupirocin 2% Nasal Ointment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Apparent Eradication of Nasal Carriage of SA
Description: Apparent eradication demonstrated by a semi-quantitative score of negative or zero using a broth enriched culture microbial assay.
Time Frame: 48 hours after the last dose of mupirocin 2%
Measure: Number; unit: participants
Arm/Group | Mupirocin 2% Nasal Ointment
Number analyzed (Participants) | 12
participants | 9

2. Secondary Outcome: The Number of Subjects With Adverse Events and Changes in Vital Signs, ECG and Routine Haematology, Clinical Chemistry and Urinalysis Tests Assessed Over the Five Day Treatment Period and Follow-up at 7 and 14 Days Relative to the First Dose.
Time Frame: 5 day treatment period and follow-up at 7 and 14 days
Measure: Number; unit: participants
Arm/Group | Mupirocin 2% Nasal Ointment
Number analyzed (Participants) | 12
participants | 0

ADVERSE EVENTS:
Arm/Group | Mupirocin 2% Nasal Ointment
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other